CLINICAL TRIAL: NCT02979873
Title: A Randomized Trial of Sirolimus (Rapamune(R)) for Relapse Prevention in Patients With Severe Aplastic Anemia Responsive to Immunosuppressive Therapy
Brief Title: Sirolimus (Rapamune ) for Relapse Prevention in People With Severe Aplastic Anemia Responsive to Immunosuppressive Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170019; 17-H-0019
Record Dates: First submitted 2016-12-01; First posted 2016-12-02 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-06

CONDITIONS: Severe Aplastic Anemia
Keywords: Rapamycin; Relapse Prevention; Immune Tolerance
MeSH Terms: conditions — Anemia, Aplastic | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirolimus (Experimental): sirolimus
  Interventions: Drug: Sirolimus
- Standard of Care (No Intervention): no intervention

INTERVENTIONS:
Drug: Sirolimus — Sirolimus will be started on day 1 for subjects in the Sirolimus arm. A baseline CBC will be obtained within one week of randomization, or on Day 0. Thereafter, CBC will be monitored on a weekly basis for subjects in both arms. In the event of relapse (see definition of outcomes Section 6.7), the patient shall return to the NIH CRC for evaluation to include bone marrow biopsy and aspirate to exclude clonal evolution to MDS. Assessment will include (i) flow cytometry phenotyping of peripheral blood mononuclear cells for regulatory T-cells (Tregs, e.g. CD4+ CD25high FOXP3+) and regulatory dendritic cells (DCregs) and (ii) proteomics assay (research labs).
  Arms: Sirolimus

SUMMARY:
Background:

People with severe aplastic anemia (SAA) do not make enough red and white blood cells, and/or platelets. Their body's immune system stops the bone marrow from making these cells. The treatment cyclosporine leads to better blood counts. But when this treatment is stopped, the disease may return in 1 in 3 people. The drug sirolimus may help by suppressing the immune system.

Objective:

To evaluate and compare the usefulness of sirolimus in preventing aplastic anemia from returning after cyclosporine is stopped, compared with stopping cyclosporine alone.

Eligibility:

People ages 2 and older with SAA who:

Have responded to immunosuppressive therapy that includes cyclosporine, and continue to take cyclosporine

Are not taking drugs with hematologic effects

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Bone marrow biopsy: The area above the hipbone will be numbed. A thin needle will remove

some bone marrow.

Participants will be randomly assigned to a group. All will stop cyclosporine. Group 1 will take sirolimus by mouth at the same time each day for 3 months with close monitoring. Group 2 will not receive the study drug but will be monitored closely.

Participants will have clinical tests for the first 3 months:

Weekly blood test

Monthly fasting blood test

For group 1, measurements of sirolimus in the blood every 1 2 weeks

Participants will have clinic visits at 3 months, 12 months, and annually for 5 years after the study starts. They may have another visit if their SAA returns. These will include:

Blood and urine tests

Bone marrow biopsy

DETAILED DESCRIPTION:
* Most acquired aplastic anemia ensues from immune-mediated destruction of hematopoietic stem and progenitor cells.
* Immunosuppression is the definitive treatment of patients with acquired aplastic anemia who are not candidates for immediate hematopoietic stem cell transplantation.
* Horse ATG combined with the calcineurin inhibitor, cyclosporine (CsA), remains standard as first-line immunosuppressive therapy (IST).
* Hematologic responses to transfusion independence occur in about two thirds of patients with standard IST and in 80-90% of patients treated with IST in combination with the growth factor eltrombopag.
* About 30% to 40% of patients relapse after discontinuation of cyclosporine.Many achieve disease control after the reinitiation of CSA, but remain CSA dependent indefinitely.
* Evidence from mouse models of bone marrow failure indicates that conversion from cyclosporine to the mTOR inhibitor, sirolimus (SRL), results in immune tolerance which can endure the eventual withdrawal of SRL.
* We hypothesize that CSA to SRL conversion will significantly decrease the relapse rate after immunosuppressive therapy for acquired aplastic anemia.
* This study will investigate the safety and efficacy of SRL for preventing relapse in patients -previously treated with IST who remain on CSA. The primary endpoint is rate of relapse at 2 years following conversion from CSA to SRL, versus stopping CSA.
* Biological sampling of peripheral blood and bone marrow aspirates during treatment will be used to investigate changes to lymphocyte phenotypes and cytokine profiles.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 2 years old
  2. Weight greater than 12 kg
  3. Previous diagnosis of SAA by bone marrow biopsy and cytogenetics, treated with lymphodepleting therapy ATG, cyclophosphamide or alemtuzumab that included cyclosporine. The lymphodepleting therapy must have been administered at least 12 months prior.
  4. Continuous treatment with cyclosporine for the previous 6 months (excluding minor dose delays not exceeding more than 30 days).
  5. Evidence of a hematologic response to an lymphodepletion-based regimen as evidence of at least two of the following:
* Absolute neutrophil count greater than or equal to 500/uL
* Platelet count greater than or equal to 20,000/uL (without transfusion support)
* Absolute reticulocyte count greater than or equal to 60,000/uL (or hemoglobin 10 gm/dL without transfusion support)

EXCLUSION CRITERIA:

1. Evidence of relapse of aplastic anemia due to cyclosporine withdrawal during the previous 6 months
2. Prior use of sirolimus or other mTOR inhibitor within 12 weeks of study entry
3. Myelodysplastic syndrome or acute myeloid leukemia, according to WHO diagnostic criteria (if baseline BM consistent with MDS after enrollment, patients will be considered ineligible and immediately exit the study, and the subject can be replaced with another subject)
4. Patients that are on CYP3A4 inhibitors and cannot replace these medications with other equivalent medications for the period of study: protease inhibitors (ritonavir, indinavir, nelfinavir, saquinavir), some macrolide antibiotics (clarithromycin, telithromycin, erythromycin), azole anti-fungals (fluconazole, itraconazole, ketoconazole), metroclopramide, felodipine, nifedipine, carbamazepine, phenobarbital, grapefruit juice and St. John s Wort.
5. Anaphylactic or hypersensitivity reaction to sirolimus
6. Patients with infections not adequately responding to appropriate therapy as evidenced by persistence of a clear source of infection that, in the view of the investigator, would preclude safe treatment with sirolimus.
7. Current pregnancy, or unwillingness to take oral contraceptives or use the barrier methods of birth control or practice abstinence to refrain from pregnancy if of childbearing potential during the course of the study 8. Lactating women, due to the potentially harmful effects on the nursing child.

9. Patients who have received live vaccines within the past 30 days

10. Patients with cancer who are actively receiving chemotherapeutic treatment or who take drugs with hematological effects such as thrombopoietin receptor agonists (such as eltrombopag), granulocyte-colony stimulating factor or erythroid stimulating agents.

11. Moribund status such that death within 7 to 10 days is likely. Comorbidities of such severity that in the view of the Investigator it would likely preclude the patient's ability to tolerate sirolimus.

12. Inability to understand the investigational nature of the study or to give informed consent or without a legally authorized representative or surrogate that can provide informed consent.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine if the rate of relapse at 24 months after CSA discontinuation can be improved by conversion to sirolimus in severe aplastic anemia patients who have responded to IST. | 24 months
  Rate of relapse in both arms

SECONDARY OUTCOMES:
Safety and tolerability of sirolimus. | 3 mo

CONTACTS AND LOCATIONS:
Overall Officials: Bhavisha A Patel, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a new requirement and the sharing of IPD is not discussed in the protocol.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0019.html